CLINICAL TRIAL: NCT04059328
Title: Use of Novel Surgical Checklists for Gynecologic Laparoscopy in Haiti: Utility in Bending the Learning Curve for Global Programs
Brief Title: Novel Surgical Checklists for Gynecologic Laparoscopy in Haiti
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Lara Harvey, Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: 181435
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Gynecology; Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physicians in Haiti: 7 OBGYN physicians underwent a laparoscopic training and simulation course and then were proctored as they performed 3 in vivo cases using a check list to help the participants remember all the steps of laparoscopic set-up.
  Interventions: Procedure: Surgical training

INTERVENTIONS:
Procedure: Surgical training — This was a gyn laparoscopy training and simulation course

SUMMARY:
The researchers traveled to University Hospital Mirebalais in Haiti and provided a one week long laparoscopic training and simulation course to the 7 OBGYN faculty there. The researchers used novel checklists to help the faculty to set up for laparoscopic cases and care for the equipment needed. The researchers then asked the physicians their opinion of the checklists.

ELIGIBILITY:
Inclusion Criteria:

* OBGYN physician in Haiti

Exclusion Criteria:

* none

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: OBGYN attendings and residents practicing at University Hospital of Mirebalais
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-09-29 (Actual); Primary Completion 2018-10-06 (Actual); Study Completion 2018-10-06 (Actual)

PRIMARY OUTCOMES:
Number of physicians that reported favoring the checklist greater than 3 on a likert scale of 1-5. | 1 week
  Likert scale 1-5. 5 indicates highest satisfaction with the checklist.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Harvey, MD MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- University Hospital at Mirebalais, Mirebalais, Haiti

IPD SHARING:
Plan to Share IPD: No